CLINICAL TRIAL: NCT01475669
Title: REPLACE (Randomized Evaluation of Fibrinogen Versus Placebo in Complex Cardiovascular Surgery): a Prospective, Multinational, Multicenter, Randomized, Double-blind, Placebo-controlled, Phase III Study for the Use of Fibrinogen Concentrate (Human) (FCH) in Complex Cardiovascular Surgery
Brief Title: Study of Fibrinogen Concentrate (Human) (FCH) to Control Bleeding During Complex Cardiovascular Surgery
Acronym: REPLACE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BI3023_3002; 2011-002685-20 (EudraCT Number)
Record Dates: First submitted 2011-11-17; First posted 2011-11-21 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Surgical Blood Loss; Postoperative Blood Loss
MeSH Terms: conditions — Blood Loss, Surgical; Postoperative Hemorrhage | interventions — Fibrinogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrinogen Concentrate (Human) (Experimental)
  Interventions: Biological: Fibrinogen Concentrate (Human) (FCH)
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Fibrinogen Concentrate (Human) (FCH) — Single dose infused intravenously within 5 minutes of the completion of the measurement of the 5-minute bleeding mass; the dose is determined individually based on the measured maximum clot firmness (MCF) and subject body weight
  Arms: Fibrinogen Concentrate (Human)
Biological: Placebo — Single dose of sodium chloride solution infused intravenously within 5 minutes at a volume equivalent to that needed for FCH
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate that Fibrinogen Concentrate (Human)(FCH) can reduce the amount of donor blood products needed during complex cardiovascular surgery, and that it is safe and well tolerated. Subjects in this study will get either a FCH or placebo infusion during surgery. This will be in addition to the standard treatment, which is donor blood or blood products. Placebo does not contain any effective medicine.

The study is randomised. This means that the likelihood that subjects will get FCH or placebo is 50%. To make the comparison between FCH and placebo as fair as possible, the study is "double blind". This means that neither the subjects nor the study doctor will know if FCH or placebo is administered. If necessary, the study doctor can find out which treatment the subjects are receiving.

ELIGIBILITY:
Inclusion Criteria:

At Screening:

* Undergoing elective open surgical procedures on any part of the aorta requiring cardiopulmonary bypass (CPB), with or without other cardiac surgical procedures (e.g. valve replacement or repair, coronary artery bypass grafting, etc.).
* 18 years of age or older.
* Written informed consent for study participation obtained before undergoing any study specific procedures.

Intraoperative (at the 1st 5-minute bleeding mass):

* A 5-minute bleeding mass of 60 to 250 g following discontinuation of CPB, administration of protamine, and establishment of surgical hemostasis.
* Minimum core body temperature 35°C, measured according to local practice.
* Activated clotting time ± 25% of baseline levels.
* Blood pH > 7.3.

Exclusion Criteria:

At Screening and/or baseline:

* Undergoing emergency aortic repair surgery.
* Reoperative aortic surgery at the same anatomic site as the original procedure such as replacement of a previously placed aortic graft. Resternotomy and rethoracotomy are permitted.
* Any operation for infection.
* Proof or suspicion of a congenital or acquired coagulation disorder (e.g. Von Willebrand's disease, hemophilia or severe liver disease) or a prothrombotic disorder (e.g. protein C or S deficiency).
* Myocardial infarction (MI), acute coronary syndrome or stroke in the 2 months preceding study surgery.
* Low molecular weight or unfractionated heparin in the 24 hours preceding study surgery.
* Clopidogrel administration within 5 days preceding study surgery or prasugrel administration within 7 days preceding study surgery or ticagrelor administration in the 48 hours preceding study surgery.
* Factor Xa inhibitors within 2 days preceding study surgery.
* IIb/IIIa antagonist administration in the 24 hours preceding study surgery.
* Use of direct thrombin inhibitors: within 3 days preceding study surgery for dabigatran and within 24 hours preceding study surgery for all others.
* An international normalized ratio > 1.3 immediately preceding the start of surgery.

Intraoperative (at the 1st 5-minute bleeding mass):

* Use of any systemic hemostatic therapy (such as FFP, platelets, prothrombin complex concentrates) from the beginning of surgery until IMP administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Total units of allogeneic blood products | Up to 24 hours after investigational medicinal product (IMP) administration
  Number of units administered of all allogeneic blood products combined (fresh frozen plasma, platelets, and red blood cells)

SECONDARY OUTCOMES:
Total avoidance of allogeneic blood transfusions | 24 hours after IMP administration
  Number of subjects who are alive and do not have any administration of platelets, fresh frozen plasma (FFP), and red blood cells (RBCs) during the first 24 hours after administration of IMP
Quantity of blood loss (6 hours) | 6 hours after skin closure
  Blood drainage volume from the chest
Quantity of blood loss (12 hours) | 12 hours after skin closure
  Blood drainage volume from the chest
Quantity of blood loss (24 hours) | 24 hours after skin closure
  Blood drainage volume from the chest
Change in bleeding mass | Immediately before and 5 minutes after completion of IMP administration
  The 5-minute bleeding mass is measured as the difference in weight of surgical swabs after 5 minutes of surgical packing of the aortic surgical site.
Mortality (Day 10) | Up to 10 days after surgery
  Mortality with adjudicated cause of death up to 10 days after surgery
Mortality (Day 30) | Up to 30 days after surgery
  Mortality with adjudicated cause of death up to 30 days after surgery
FFP consumption (24 hours) | 24 hours after IMP administration
FFP consumption (10 days) | 10 days after IMP administration
Platelet consumption (24 hours) | 24 hours after IMP administration
Platelet consumption (10 days) | 10 days after IMP administration
Red blood cells (RBC) consumption (24 hours) | 24 hours after IMP administration
RBC consumption (10 days) | 10 days after IMP administration
Total units of all allogeneic blood products (6 hours) | 6 hours after IMP administration
  Number of units of all allogeneic blood products combined (FFP, platelets, and/or RBCs) administered during the first 6 hours after administration of IMP
Total units of all allogeneic blood products (12 hours) | 12 hours after IMP administration
  Number of units of all allogeneic blood products combined (FFP, platelets, and/or RBCs) administered during the first 12 hours after administration of IMP
Volume of all allogeneic blood products (6 hours) | 6 hours after IMP administration
  Volume of all allogeneic blood products combined (FFP, platelets, and/or RBCs) administered during the first 6 hours after administration of IMP
Volume of all allogeneic blood products (12 hours) | 12 hours after IMP administration
  Volume of all allogeneic blood products combined (FFP, platelets, and/or RBCs) administered during the first 12 hours after administration of IMP
Volume of all allogeneic blood products (24 hours) | 24 hours after IMP administration
  Volume of all allogeneic blood products combined (FFP, platelets, and/or RBCs) administered during the first 24 hours after administration of IMP
Time from administration of study drug to completion of skin closure | Average 2 hours
Mortality (24 hours) | WIthin 24 hours after IMP administration
  Mortality with adjudicated cause of death during the first 24 hours after administration of IMP
Peak plasma concentration of fibrinogen (Cmax) | At up to 10 time points from baseline and up to Day 11 after surgery.
Maximum clot firmness | At baseline; on the day of surgery at: 30 min before CPB, the 1st 5 min bleeding mass, the end of IMP infusion, the 2nd 5-min bleeding mass, and closure; and on Day 2, 3, 4 and at the end of the study (discharge/Day 11 or at discontinuation if earlier).

CONTACTS AND LOCATIONS:
Overall Officials: Niels Rahe-Meyer, MD, PhD, Principal Investigator — Hannover Medical School
Locations (35):
- Allgemeines Krankenhaus der Stadt Wien - Universitätskliniken, Vienna, Austria
- Brazil (2):
  - Fundacao Universitaria de Cardiologia - Instituto de Cardiol, Porto Alegre, Rio Grande do Sul
  - InCor, São Paulo, São Paulo
- Canada (6):
  - Providence Health-St Paul's Hospital, Vancouver, British Columbia
  - Hamilton Health Science, Hamilton, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - University of Toronto - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Universite Laval - Cardiologie et de Pneumologie de Quebec, Sainte-Foy, Quebec
- Czechia (2):
  - University Hospital St. Anna Brno, Brno
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
- Kobenhavns Universitet-Det Sundhedsvidenskabelige Fakultet, Copenhagen, Denmark
- HUCH Anaestesia and Surgery, Helsinki, Finland
- Germany (3):
  - Klinikum der Universität München, Munich, Bavaria
  - Klinikum der J.-W.-Goethe-Universität, Frankfurt am Main, Hesse
  - Study Site, Bielefeld/Hannover
- Italy (3):
  - Policlinico S. Orsola Malpighi, Bologna
  - Fondazione Centro San Raffaele, Milan
  - Azienda Ospedaliera di Udine, Udine
- Japan (9):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Kurume University Hospital, Kurume, Fukuoka
  - Hamamatsu University Hospital, Hamamatsu, Higashi-ku
  - Kobe University Hospital, Kobe, Hyōgo
  - Kyoto University Hospital, Kyoto, Kamigyo-ku
  - Tohoku University Hospital, Sendai, Miyagi
  - Tenri Hospital, Tenri, Nara
  - National Cerebral and Cardiovascular Center, Suita, Osaka, Osaka
  - Keio University Hospital, Shinjuku
- Poland (3):
  - Inst. Kardiologii im. Prymasa Tysiaclecia Kard. S. Wyszynskiego, Warszawa - Anin, Masovian Voivodeship
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Samodzielny Publiczny Szpital Kliniczny nr 2, Szczecin
- United Kingdom (4):
  - Papworth Hospital, Cambridge
  - University Hospital of Leicester, Leicester
  - Liverpool Heart and Chest Hospital, Liverpool
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Rahe-Meyer N, Levy JH, Mazer CD, Schramko A, Klein AA, Brat R, Okita Y, Ueda Y, Schmidt DS, Gill R. Randomized evaluation of fibrinogen versus placebo in complex cardiovascular surgery: post hoc analysis and interpretation of phase III results. Interact Cardiovasc Thorac Surg. 2019 Apr 1;28(4):566-574. doi: 10.1093/icvts/ivy302. PMID 30462259
- [Derived] Rahe-Meyer N, Levy JH, Mazer CD, Schramko A, Klein AA, Brat R, Okita Y, Ueda Y, Schmidt DS, Ranganath R, Gill R. Randomized evaluation of fibrinogen vs placebo in complex cardiovascular surgery (REPLACE): a double-blind phase III study of haemostatic therapy. Br J Anaesth. 2016 Jul;117(1):41-51. doi: 10.1093/bja/aew169. PMID 27317703